CLINICAL TRIAL: NCT03224572
Title: The Effect of Vitamin C on Quality of Life of Terminal Cancer Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201702008MIPB
Record Dates: First submitted 2017-07-16; First posted 2017-07-21 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-04

CONDITIONS: Vitamin C Deficiency
Keywords: vitamin C; quality of life; terminal cancer
MeSH Terms: conditions — Ascorbic Acid Deficiency | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Randomized double-blinded controlled trial
Who Masked: Participant, Care Provider
Masking Description: double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The study group (Experimental): The study group will receive intravenous high-dose vitamin C 30 gm in 500 ml normal saline in 1-hour infusion, once per week, and total 4-week treatment.
  Interventions: Drug: high-dose vitamin C 30gm; Other: normal saline
- The control group (Placebo Comparator): The control group will receive 500 ml normal saline in 1-hour infusion, once per week, and total 4-week treatment.
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: high-dose vitamin C 30gm — High-dose vitamin C 30 gm in 500 ml normal saline, once per week, and total 4-week treatment.
  Other Names: ascorbic acid 30 gm
  Arms: The study group
Other: normal saline — 500ml normal saline, once per week, and total 4-week treatment

SUMMARY:
This study determines whether high dose vitamin C is effective for quality of life in terminal cancer patients.

DETAILED DESCRIPTION:
The investigator's project is a single medical center, randomized double- blinded trial. The target group is terminal cancer patients at Palliative care clinics. The experimental group will receive intravenous high-dose vitamin C 30 g in 500 ml normal saline in 1-hour infusion, once per week, and total 4-week treatment. The control group will receive 500 ml normal saline in 1-hour infusion, once per week, and total 4-week treatment. The primary outcome is the improvement of quality of life, measured by European Organization for Research and Treatment of cancer (EORTC). The secondary outcome is the survival analysis.The participants will be followed up weekly for 2 weeks, then bi-weekly for 6 months.

ELIGIBILITY:
Inclusion Criteria:

-Terminal colon cancer patients without pleural effusions, who will not receive any curative radiotherapy or chemotherapy.

Exclusion Criteria:

* Renal metastasis or obstructive uropathy by radiology
* Nephrotic syndrome
* Creatinine over 1.5mg/dl
* Urolithasis
* Under other folk therapy or vitamin infusion therapy
* Those who can't exercise the right of consent
* Those who can't answer the questionaires
* Glucose-6-Phosphate Dehydrogenase Deficiency
* Severe lower leg edema or general edema

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The improvement of quality of life (QOL) | 6 months
  QOL measured by European Organization for Research and Treatment of cancer Quality of Life Questionnaire (EORTC QLQ)-C30

SECONDARY OUTCOMES:
Survival analysis | 6 months
  death time of those who have completed the 4-week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Ying Chen, MD, MHSc, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No